CLINICAL TRIAL: NCT05296863
Title: Adipose-derived Stem Cell Conditioned Media as a Novel Approach for Hair Regrowth in Male Androgenetic Alopecia: A Randomized, Double-blind Clinical Trial
Brief Title: Adipose-derived Stem Cell Conditioned Media as a Novel Approach for Hair Regrowth in Male Androgenetic Alopecia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. dr. Lili Legiawati, SpKK(K) (Other)
Collaborators: Kementerian Riset dan Teknologi / Badan Riset dan Inovasi Nasional, Indonesia (Other Government); PT. Kimia Farma (Persero) Tbk (Industry)
Responsible Party: Sponsor-Investigator, Dr. dr. Lili Legiawati, SpKK(K), Principal Investigator, Indonesia University
Organization: Indonesia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KET-19UN2.F1ETIKPPM00022020
Record Dates: First submitted 2022-02-18; First posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Alopecia, Androgenetic; Hair Loss/Baldness
Keywords: Stem cell therapy; Adipose derived stem cell conditioned media; Hair regeneration
MeSH Terms: conditions — Alopecia | interventions — Minoxidil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-concentrated ADSC-CM (Experimental): 2 ml intradermal injection of non-concentrated ADSC-CM + 1 ml of 5% topical Minoxidil daily
  Interventions: Combination Product: Non-concentrated adipose-derived stem cell conditioned media and 5% Minoxidil; Combination Product: Placebo and 5% Minoxidil
- Concentrated ADSC-CM (Experimental): 2 ml intradermal injection of concentrated ADSC-CM + 1 ml of 5% topical Minoxidil daily
  Interventions: Combination Product: Concentrated adipose-derived stem cell conditioned media and 5% Minoxidil; Combination Product: Placebo and 5% Minoxidil

INTERVENTIONS:
Combination Product: Non-concentrated adipose-derived stem cell conditioned media and 5% Minoxidil — Non-concentrated ADSC-CM is given during week 0, 2, 4, and 6 on the left side of the scalp.
  Minoxidil is applied twice using a spray, in the morning and at night.
  Arms: Non-concentrated ADSC-CM
Combination Product: Concentrated adipose-derived stem cell conditioned media and 5% Minoxidil — Intervention is given during week 0, 2, 4, and 6 on the left side of the scalp. Minoxidil is applied twice using a spray, in the morning and at night.
  Arms: Concentrated ADSC-CM
Combination Product: Placebo and 5% Minoxidil — Intervention is given during week 0, 2, 4, and 6 on the right side of the scalp.
  Minoxidil is applied twice using a spray, in the morning and at night.

SUMMARY:
This study investigated the efficacy of adipose derived stem cell conditioned media (ADSC-CM) combined with minoxidil for hair regeneration therapy in male AGA.

DETAILED DESCRIPTION:
This study was a double-blind, randomized clinical trial (RCT). Two concentrations of ADSC-CM were utilized: concentrated and non-concentrated ADSC-CM. The scalp was divided vertically in half; one side was injected with 2 ml of ADSC-CM, while the control side received 2 ml of NaCl 0,9%. After the injection, patients applied topical 5% minoxidil twice daily. Clinical improvements were assessed using photographic evaluation and trichoscan every two weeks.

ELIGIBILITY:
Inclusion Criteria:

* males aged 25-58 years old
* Hamilton-Norwood criteria grades II to VI
* cessation of anti-androgens and minoxidil treatment for at least one month

Exclusion Criteria:

* patients with hair loss other than AGA, such as alopecia areata, chemotherapy-induced alopecia, autoimmune-induced alopecia, and scalp malignancies;
* patients receiving 5-alpha reductase inhibitor therapy;
* patients who had received growth factor treatment (platelet-rich plasma or microneedling) for at least six months prior to the study; and
* history of hypertrophic scars or blood clotting disorders.

Ages: 25 Years to 58 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Hair count | Within 6 weeks
  Sum of hair
Hair density | Within 6 weeks
  count/cm2
Terminal rate | Within 6 weeks
  Percentage of terminal hairs
Vellus rate | Within 6 weeks
  Percentage of terminal hairs
Mean thickness | Within 6 weeks
  In centimeters
Total follicular units | Within 6 weeks
  Unit of hair follicles

SECONDARY OUTCOMES:
7-point scale | Within 6 weeks
  In order to assess patient satisfaction of the research process and treatment outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Universitas Indonesia, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

REFERENCES:
- [Background] Al Aboud AM, Syed HA, Zito PM. Alopecia. 2024 Feb 26. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK538178/ PMID 30844205
- [Background] Salman KE, Altunay IK, Kucukunal NA, Cerman AA. Frequency, severity and related factors of androgenetic alopecia in dermatology outpatient clinic: hospital-based cross-sectional study in Turkey. An Bras Dermatol. 2017 Jan-Feb;92(1):35-40. doi: 10.1590/abd1806-4841.20175241. PMID 28225954
- [Background] Nestor MS, Ablon G, Gade A, Han H, Fischer DL. Treatment options for androgenetic alopecia: Efficacy, side effects, compliance, financial considerations, and ethics. J Cosmet Dermatol. 2021 Dec;20(12):3759-3781. doi: 10.1111/jocd.14537. Epub 2021 Nov 6. PMID 34741573
- [Background] Huang CH, Fu Y, Chi CC. Health-Related Quality of Life, Depression, and Self-esteem in Patients With Androgenetic Alopecia: A Systematic Review and Meta-analysis. JAMA Dermatol. 2021 Aug 1;157(8):963-970. doi: 10.1001/jamadermatol.2021.2196. PMID 34232264
- [Background] Varothai S, Bergfeld WF. Androgenetic alopecia: an evidence-based treatment update. Am J Clin Dermatol. 2014 Jul;15(3):217-30. doi: 10.1007/s40257-014-0077-5. PMID 24848508
- [Background] Ferreira JR, Teixeira GQ, Santos SG, Barbosa MA, Almeida-Porada G, Goncalves RM. Mesenchymal Stromal Cell Secretome: Influencing Therapeutic Potential by Cellular Pre-conditioning. Front Immunol. 2018 Dec 4;9:2837. doi: 10.3389/fimmu.2018.02837. eCollection 2018. PMID 30564236
- [Background] Khandpur S, Gupta S, Gunaabalaji DR. Stem cell therapy in dermatology. Indian J Dermatol Venereol Leprol. 2021 Nov-Dec;87(6):753-767. doi: 10.25259/IJDVL_19_20. PMID 34245532
- [Background] Owczarczyk-Saczonek A, Wocior A, Placek W, Maksymowicz W, Wojtkiewicz J. The Use of Adipose-Derived Stem Cells in Selected Skin Diseases (Vitiligo, Alopecia, and Nonhealing Wounds). Stem Cells Int. 2017;2017:4740709. doi: 10.1155/2017/4740709. Epub 2017 Aug 21. PMID 28904532
- [Background] Tsuji W, Rubin JP, Marra KG. Adipose-derived stem cells: Implications in tissue regeneration. World J Stem Cells. 2014 Jul 26;6(3):312-21. doi: 10.4252/wjsc.v6.i3.312. PMID 25126381
- [Background] Kim WS, Park BS, Sung JH, Yang JM, Park SB, Kwak SJ, Park JS. Wound healing effect of adipose-derived stem cells: a critical role of secretory factors on human dermal fibroblasts. J Dermatol Sci. 2007 Oct;48(1):15-24. doi: 10.1016/j.jdermsci.2007.05.018. Epub 2007 Jul 23. PMID 17643966
- [Background] Fukuoka H, Suga H. Hair Regeneration Treatment Using Adipose-Derived Stem Cell Conditioned Medium: Follow-up With Trichograms. Eplasty. 2015 Mar 26;15:e10. eCollection 2015. PMID 25834689
- [Background] Shin H, Ryu HH, Kwon O, Park BS, Jo SJ. Clinical use of conditioned media of adipose tissue-derived stem cells in female pattern hair loss: a retrospective case series study. Int J Dermatol. 2015 Jun;54(6):730-5. doi: 10.1111/ijd.12650. Epub 2015 Mar 16. PMID 25777970
- [Background] Narita K, Fukuoka H, Sekiyama T, Suga H, Harii K. Sequential Scalp Assessment in Hair Regeneration Therapy Using an Adipose-Derived Stem Cell-Conditioned Medium. Dermatol Surg. 2020 Jun;46(6):819-825. doi: 10.1097/DSS.0000000000002128. PMID 31490301
- [Background] Lee SB, Shin HT, Byun JW, Shin J, Choi GS. Clinical efficacy of adipocyte-derived stem cells conditioned media combined with micro-injury in refractory patch of alopecia areata. Arch Dermatol Res. 2022 Aug;314(6):527-532. doi: 10.1007/s00403-021-02252-9. Epub 2021 Jun 15. PMID 34131795
- [Background] Tak YJ, Lee SY, Cho AR, Kim YS. A randomized, double-blind, vehicle-controlled clinical study of hair regeneration using adipose-derived stem cell constituent extract in androgenetic alopecia. Stem Cells Transl Med. 2020 Aug;9(8):839-849. doi: 10.1002/sctm.19-0410. Epub 2020 May 18. PMID 32420695
- [Background] Gupta AK, Quinlan EM, Venkataraman M, Bamimore MA. Microneedling for Hair Loss. J Cosmet Dermatol. 2022 Jan;21(1):108-117. doi: 10.1111/jocd.14525. Epub 2021 Oct 29. PMID 34714971
- [Background] Kumar MK, Inamadar AC, Palit A. A Randomized Controlled, Single-Observer Blinded Study to Determine the Efficacy of Topical Minoxidil plus Microneedling versus Topical Minoxidil Alone in the Treatment of Androgenetic Alopecia. J Cutan Aesthet Surg. 2018 Oct-Dec;11(4):211-216. doi: 10.4103/JCAS.JCAS_130_17. PMID 30886475
- [Background] Gajjar PC, Mehta HH, Barvaliya M, Sonagra B. Comparative Study between Mesotherapy and Topical 5% Minoxidil by Dermoscopic Evaluation for Androgenic Alopecia in Male: A Randomized Controlled Trial. Int J Trichology. 2019 Mar-Apr;11(2):58-67. doi: 10.4103/ijt.ijt_89_18. PMID 31007474
- [Background] York K, Meah N, Bhoyrul B, Sinclair R. A review of the treatment of male pattern hair loss. Expert Opin Pharmacother. 2020 Apr;21(5):603-612. doi: 10.1080/14656566.2020.1721463. Epub 2020 Feb 17. PMID 32066284
- [Background] Rossi A, Anzalone A, Fortuna MC, Caro G, Garelli V, Pranteda G, Carlesimo M. Multi-therapies in androgenetic alopecia: review and clinical experiences. Dermatol Ther. 2016 Nov;29(6):424-432. doi: 10.1111/dth.12390. Epub 2016 Jul 18. PMID 27424565
- [Background] Krupa Shankar D, Chakravarthi M, Shilpakar R. Male androgenetic alopecia: population-based study in 1,005 subjects. Int J Trichology. 2009 Jul;1(2):131-3. doi: 10.4103/0974-7753.58556. PMID 20927235
- [Background] Ding Q, Xu YX, Sun WL, Liu JJ, Deng YY, Wu QF, Cao CY, Zhou LB, Lu Y, Fan WX. Early-onset androgenetic alopecia in China: a descriptive study of a large outpatient cohort. J Int Med Res. 2020 Mar;48(3):300060519897190. doi: 10.1177/0300060519897190. PMID 32188323
- [Background] Banger HS, Malhotra SK, Singh S, Mahajan M. Is Early Onset Androgenic Alopecia a Marker of Metabolic Syndrome and Carotid Artery Atherosclerosis in Young Indian Male Patients? Int J Trichology. 2015 Oct-Dec;7(4):141-7. doi: 10.4103/0974-7753.171566. PMID 26903742
- [Background] Arias-Santiago S, Gutierrez-Salmeron MT, Buendia-Eisman A, Giron-Prieto MS, Naranjo-Sintes R. A comparative study of dyslipidaemia in men and woman with androgenic alopecia. Acta Derm Venereol. 2010 Sep;90(5):485-7. doi: 10.2340/00015555-0926. PMID 20814623
- [Background] Kim MW, Shin IS, Yoon HS, Cho S, Park HS. Lipid profile in patients with androgenetic alopecia: a meta-analysis. J Eur Acad Dermatol Venereol. 2017 Jun;31(6):942-951. doi: 10.1111/jdv.14000. Epub 2016 Nov 2. PMID 27717019
- [Background] Won CH, Park GH, Wu X, Tran TN, Park KY, Park BS, Kim DY, Kwon O, Kim KH. The Basic Mechanism of Hair Growth Stimulation by Adipose-derived Stem Cells and Their Secretory Factors. Curr Stem Cell Res Ther. 2017;12(7):535-543. doi: 10.2174/1574888X12666170829161058. PMID 28875863
- [Background] Fabbrocini G, Fardella N, Monfrecola A, Proietti I, Innocenzi D. Acne scarring treatment using skin needling. Clin Exp Dermatol. 2009 Dec;34(8):874-9. doi: 10.1111/j.1365-2230.2009.03291.x. Epub 2009 May 22. PMID 19486041
- [Background] Ramdasi S, Tiwari SK. Human Mesenchymal Stem Cell-Derived Conditioned Media for Hair Regeneration Applications. J Stem Cells. 2016;11(4):201-211. PMID 28296872
- [Background] Xiao S, Deng Y, Mo X, Liu Z, Wang D, Deng C, Wei Z. Promotion of Hair Growth by Conditioned Medium from Extracellular Matrix/Stromal Vascular Fraction Gel in C57BL/6 Mice. Stem Cells Int. 2020 Jun 13;2020:9054514. doi: 10.1155/2020/9054514. eCollection 2020. PMID 32612663
- [Background] Mecklenburg L, Tobin DJ, Muller-Rover S, Handjiski B, Wendt G, Peters EM, Pohl S, Moll I, Paus R. Active hair growth (anagen) is associated with angiogenesis. J Invest Dermatol. 2000 May;114(5):909-16. doi: 10.1046/j.1523-1747.2000.00954.x. PMID 10771470
- [Derived] Legiawati L, Suseno LS, Sitohang IBS, Yusharyahya SN, Pawitan JA, Liem IK, Kurniawati T, Ardelia A, Paramastri K. Combination of adipose-derived stem cell conditioned media and minoxidil for hair regrowth in male androgenetic alopecia: a randomized, double-blind clinical trial. Stem Cell Res Ther. 2023 Aug 21;14(1):210. doi: 10.1186/s13287-023-03440-2. PMID 37605227